CLINICAL TRIAL: NCT00450970
Title: Expanded Access Study of Satraplatin Plus Prednisone in Patients With Hormone Refractory Prostate Cancer (HRPC) Previously Treated With Unlimited Cytotoxic Chemotherapy Regimen (SPERA)
Brief Title: Expanded Access Study of Satraplatin Plus Prednisone in Patients With Hormone Refractory Prostate Cancer (HRPC)
Acronym: SPERA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decided to discontinue study drug development.
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAT3-06-04
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Prostate Cancer
Keywords: Hormone Refractory Prostate Cancer (HRPC); Hormone Refractory Prostate Cancer; Unlimited Prior Cytotoxic Chemotherapy Regimens
MeSH Terms: conditions — Prostatic Neoplasms | interventions — satraplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Prednisone and Satraplatin (INN / USAN), also known as JM-216, or OC-6-43-bis(acetato-O)ammine dichloro (cyclohexanamine)-platinum (IV), is a member of a novel class of platinum (IV) compounds that are absorbed by the oral route. The lipophilic properties of these compounds, and hence their absorption, are largely determined by the nature of the axial acetate ligands.
  Interventions: Drug: Oral Satraplatin
- 2 (Experimental): Prednisone (17 alpha, 21-dihydroxypregna-1, 4-diene-3, 11, 20-trione) is commercially formulated as the acetate salt (prednisone 21-acetate). It is a biologically inert glucocorticoid, which is converted to active prednisolone in the liver.
  Interventions: Drug: Oral Satraplatin

INTERVENTIONS:
Drug: Oral Satraplatin — The SPERA protocol states that satraplatin may be continued until evidence of disease progression (at the discretion of the investigator), intolerable toxicity, withdrawal of informed consent, or non compliance. The treatment consists of satraplatin 80 mg/m2 administered by mouth once daily for five consecutive days (days 1-5) plus prednison 5 mg po twice daily. The treatment cycle is repeated every 35 days.

SUMMARY:
The SPERA trial is designed to 1. provide satraplatin to physicians with patients who have hormone refractory prostate cancer (HRPC) which has progressed following unlimited cytotoxic chemotherapy regimens for metastatic disease and 2. to evaluate the safety of oral satraplatin in this patient population.

DETAILED DESCRIPTION:
*****UPDATE***** On October 30th, 2007 GPC Biotech announced topline overall survival results for the Phase III trial in hormone refractory prostate cancer-Satraplatin and Prednisone Against Refractory Cancer (SPARC) trial.

The trial evaluated satraplatin plus prednisone versus placebo plus prednisone as a second-line treatment in 950 patients with hormone-refractory prostate cancer (HRPC). The companies reported that the trial did not achieve the endpoint of overall survival (p=0.80, stratified log rank analysis). The median was 61.3 weeks for the satraplatin arm compared to 61.4 weeks for the control group and the hazard ratio was 0.97 (95% CI: 0.83, 1.13). The companies are currently conducting pre-specified subset analyses.

Satraplatin is a member of the platinum-based class of chemotherapy drugs. Platinum-based drugs have been clinically proven to be one of the most effective classes of anticancer therapies. Unlike the currently marketed platinum-based drugs, satraplatin can be given orally.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic(Stage D2)prostate cancer
* Progression after unlimited prior cytotoxic chemotherapy regimens
* ECOG Performance status equal/less than 2
* Surgical or medical castration
* Adequate bone marrow, liver, and renal function
* Informed consent
* Patients treated with bisphosphonates prior to entry are eligible and should continue bisphosphonates therapy while on this trial

Exclusion Criteria:

* Serious concurrent uncontrolled medical disorder
* Malignant disease requiring on-going therapy
* Prior significant RT/radionuclide therapy
* Major GI surgery or GI disease affecting absorption
* Disease where corticosteroids are contraindicated
* Brain metastases
* Poorly-controlled or uncontrolled insulin-dependent diabetes

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2007-02; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The SPERA trial is designed to provide satraplatin to physicians with patients who have hormone refractory prostate cancer (HRPC) which has progressed following unlimited prior cytotoxic chemotherapy regimens for metastatic disease. | Patient evaluation by MD at baseline to determine eligibility.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Pultar, MD, Study Director — GPC Biotech Inc.
Locations (121):
- United States (121):
  - Carraway Cancer Clinic, Birmingham, Alabama
  - Birmingham Hematology and Oncology, Birmingham, Alabama
  - Urology Centers of Alabama, Homewood, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Clopton Clinic, Jonesboro, Arkansas
  - Pacific Cancer Medical Center, Inc, Anaheim, California
  - East Valley Hematology Oncology Medical Group, Burbank, California
  - Pacific Shores Medical Group, Long Beach, California
  - North Valley Hematology/Oncology Medical Group, Mission Hills, California
  - Michael Harris MD, Mission Viejo, California
  - Newport Cancer Care Medical Assoc., Inc., Newport Beach, California
  - Medical Oncology Care Associates, Orange, California
  - Desert Cancer Center, Rancho Mirage, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Santa Barbara Hematology Oncology Medical Group, Santa Barbara, California
  - Santa Barbara Hemotology, Santa Barbara, California
  - Stockton Hematology Oncology Medical Group, Stockton, California
  - Sierra Nevada Oncology, Truckee, California
  - Rocky Mountain Cancer Center, Colorado Springs, Colorado
  - Oncology Associates of Bridgeport, Bridgeport, Connecticut
  - Medical Specialists of Fairfield, LLC, Fairfield, Connecticut
  - Davis, Posteraro, and Wasser, MDs, LLP, Manchester, Connecticut
  - Whittigham Cancer Center at Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Hematology Oncology, Stamford, Connecticut
  - Connecticut Oncology & Hematology, LLP, Torrington, Connecticut
  - Center for Hematology-Oncology, Boca Raton, Florida
  - Florida Cancer Specalists, Bradenton, Florida
  - Florida Cancer Care Specialists-Fort Myers Summerlin Office, Fort Myers, Florida
  - Gainesville Hematology Oncology Associates, Gainesville, Florida
  - ICON, Jacksonville, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - MIMA Century Research Assoc., Melbourne, Florida
  - Marc I. Saltzman, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Mid-Florida Hematology & Oncology Centers, Orange City, Florida
  - Sacred Heart Hospital Cancer Research, Pensacola, Florida
  - Florida Cancer Specialists, Port Charlotte, Florida
  - Notheast Georgia Cancer Care, LLC, Athens, Georgia
  - Medical Oncology Assoc. of Augusta, PC, Augusta, Georgia
  - GA Urology, Decatur, Georgia
  - Suburban Hematology-Oncology Assoc., PC, Lawrenceville, Georgia
  - University of Chicago, Chicago, Illinois
  - Medical & Surgical Spealists, LLC, Galesburg, Illinois
  - Urology Associates, S.C., Mattoon, Illinois
  - Mid-Illinois Hematology and Oncology Assoc., LTD, Normal, Illinois
  - Oncology Hematology Associates of Central IL, PC, Peoria, Illinois
  - Fort Wayne Medical Oncology Hematology, Inc., Fort Wayne, Indiana
  - Mahendra M. Shah, MD, FACP, Hammond, Indiana
  - McFarland Clinic PC, Ames, Iowa
  - Iowa Blood and Cancer Care, PLC, Cedar Rapids, Iowa
  - Heartland Oncology & Hematology, LLP, Council Bluffs, Iowa
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - Drs.Caroll, Sheth and Raghavan, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - The Center for Clinical Research, Hagerstown, Maryland
  - Associates in Oncology/Hematology, Rockville, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Kalamazoo Hematology and Oncology, Kalamazoo, Michigan
  - Jackson Oncology Associates, Jackson, Mississippi
  - NW MS Hem/Onc (Tupelo), Tupelo, Mississippi
  - Columbia Comprehensive Cancer Care Center, Columbia, Missouri
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - St. Johns Mercy Medical Center, St Louis, Missouri
  - The Center for Cancer Care & Research, St Louis, Missouri
  - The Billings Clinic, Billings, Montana
  - Saint Francis Memoiral Hospital, Grand Island, Nebraska
  - Nebraska Hematology-Oncology,PC, Lincoln, Nebraska
  - Cancer Care at St. Claire's, Denville, New Jersey
  - Hematology Oncology Associates of Northern New Jersey, Morristown, New Jersey
  - Northern Valley Medical, Westwood, New Jersey
  - Hematology Oncology Assoc. of W. Suffolk, PC, Bay Shore, New York
  - The Mary Imogene Bassett Hospital, Cooperstown, New York
  - North Shore Hematology Oncology Assoc., East Setauket, New York
  - Richmond University Medical Center, Staten Island, New York
  - Gaston Hematology and Oncology, Gastonia, North Carolina
  - Cancer Center of North Carolina, Raleigh, North Carolina
  - MeritCare Clinical Research, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Tricounty Hem/Onc Associates, Canton, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Mid-Ohio Oncology/Hematology, Columbus, Ohio
  - Hematology-Oncology Consultants, Inc, Columbus, Ohio
  - Ohio Cancer Specialists, Mansfield, Ohio
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Specialists of Oklahoma, Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Lancaster Cancer Center, Ltd., Lancaster, Pennsylvania
  - Greater Philadelphia Cancer Center, Philadelphia, Pennsylvania
  - Carolina Health Care, Florence, South Carolina
  - Mid-South Cancer Center, PC, Germantown, Tennessee
  - Mid-South Cancer Center, Germantown, Tennessee
  - The Jones Clinic, Germantown, Tennessee
  - McLeod Cancer and Blood Center, Johnson City, Tennessee
  - Kingsport Hematology Oncology, Kingsport, Tennessee
  - Boston Baskin Cancer Group D/B/A/ UTCI, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Texas Oncology Cancer Center, PA, Austin, Texas
  - Lone Star Oncology Consultants, Austin, Texas
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Mitchell Medical Clinic, Daingerfield, Texas
  - Center for Oncology Research and Treatment, Dallas, Texas
  - Texas Oncology, Dallas, Texas
  - Clinical Oncology & Hematology, LLP, Dallas, Texas
  - Dallas Oncology Consultants, PA, Dallas, Texas
  - Texas Cancer Center, Denton, Texas
  - Cancer Care Centers of South Texas, Fredericksburg, Texas
  - Allison Cancer Center, Midland, Texas
  - Cancer Care Centers of South Texas, New Braunfels, Texas
  - Northern Utah Associates, Ogden, Utah
  - Peninsula Cancer Institute, Newport News, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Sacred Heart Medical Center - Providence Cancer Care Center, Spokane, Washington
  - Northwest Cancer Specialists, PC, Vancouver, Washington
  - Green Bay Oncology, Ltd., Green Bay, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin